CLINICAL TRIAL: NCT01990846
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Assessment of the Safety, Tolerability and Pharmacokinetics of Escalating Single and Repeat Doses of Flufirvitide-3 Dry Powder for Inhalation in Healthy Subjects
Brief Title: Safety, Tolerability, and PK of Escalating Doses of Flufirvitide-3 Dry Powder for Inhalation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autoimmune Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIT02-1002
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: antiviral, influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Flufirvitide-3 dose level 1 (Experimental): Single dose administration for dose level 1
  Interventions: Drug: Flufirvitide 3
- Flufirvitide 3-Dose level 2 (Experimental): Single dose administration for Dose Level 2
  Interventions: Drug: Flufirvitide 3
- Placebo (Placebo Comparator): Single Dose administration Placebo for Flufirvitide-3
  Interventions: Drug: Placebo for Flufirvitide-3
- Flufirvitide-3 Dose level 1- Repeat dose (Experimental): Repeat dose administration for five days
  Interventions: Drug: Flufirvitide 3
- Flufirvitide-3-Dose level 2 Repeat dose (Experimental): Repeat dose administration for 5 days
  Interventions: Drug: Flufirvitide 3
- Placebo for Flufirvitide-3 Repeat dose (Placebo Comparator): Repeat dose administration for 5 days
  Interventions: Drug: Placebo for Flufirvitide-3

INTERVENTIONS:
Drug: Flufirvitide 3
  Other Names: FF-3
  Arms: Flufirvitide 3-Dose level 2; Flufirvitide-3 Dose level 1- Repeat dose; Flufirvitide-3 dose level 1; Flufirvitide-3-Dose level 2 Repeat dose
Drug: Placebo for Flufirvitide-3
  Arms: Placebo; Placebo for Flufirvitide-3 Repeat dose

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics (PK) of single,and repeat escalating doses of FF-3 dry powder administered via inhalation in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant, non-lactating female subjects of 18 to 50 years of age inclusive.
2. Body Mass Index (BMI) of 18 to 30 kg/m2 inclusive and body weight of 50 to 100 kg inclusive.
3. Normal spirometry values at Screening and Baseline defined as forced vital capacity (FVC) and forced expiratory volume in one second (FEV1) greater than 80% predicted or above the LLN and the FEV1/FVC ratio greater than 70%. Results of FEV1 and FVC must be reproducible (± 5%) between Screening and Baseline.
4. Post-menopausal women with amenorrhea for at least 2 years will be eligible (confirmed by follicle stimulating hormone [FSH] test).
5. Females of childbearing potential must use acceptable birth control methods throughout the study and for 30 days after the last dose of the IMP:
6. Male subjects:

   1. Must agree to use a condom (or diaphragm plus spermicide in female partner) from the time of the first dose of IMP through 90 days after the last dose.
   2. Must agree to not donate sperm for 90 days after the last dose of IMP.
   3. Vasectomies in males for 6 months minimum prior to the first dose of the IMP are an acceptable form of contraception.
   4. Males who claim abstinence as their method of contraception are allowed provided they agree to use a barrier method (diaphragm plus spermicide in female partner or condom) should they become sexually active from screening to 90 days after the last dose of IMP.
7. Willing and able to provide written informed consent and provide authorization for use of protected health information (HIPAA).
8. Willing and able to adhere to the lifestyle guideline restrictions outlined in the protocol.
9. Willing and able to be confined to the CRU as required by the protocol.

Exclusion Criteria

1. Evidence of or history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine, or psychiatric disease, or current clinically significant infection.
2. History and/or presence of asthma at Screening or Baseline; presence of active rhinitis or sinusitis at Screening or Baseline.
3. Clinically significant nasal abnormalities including nasal septum deviation, septum perforations, or polyps, history of recurrent epistaxis, history of sinus surgery and/or persistent hypertrophic inferior turbinates.
4. Clinically significant abnormalities at Screening or Baseline in safety laboratory tests, ECGs, or spirometry.
5. Inability to perform spirometry according to the 2005 American Thoracic Society (ATS) acceptability and repeatability standards.
6. History of significant nasal irritation from use of nasal sprays or drops.
7. Corrected QT interval (QTc) greater than 450 msec for males and 470 msec for females as corrected by the Fridericia formula.
8. History of drug or alcohol abuse within the past 2 years; current excessive user of alcohol defined as regular weekly intake of greater than 15 units for male subjects and 10 units for female subjects. One unit equals 25 mL spirits, 125 mL wine or 250 mL beer.
9. Tobacco users (includes users who stopped smoking £90 days prior to the screening evaluation). [Note: "Tobacco use" includes smoking and the use of snuff and chewing tobacco, and other nicotine or nicotine containing products.]
10. Received an IMP or participated in another research study within 30 days of the first dose of the IMP for this study.
11. Participated in a previous investigational study of FF3.
12. History of influenza vaccination with a live vaccine within 7 days or with an attenuated vaccine within 14 days of the first dose of IMP.
13. Use of prescription drugs within 14 days prior to the first dose of IMP, excepting oral contraceptives.
14. Received any non-prescription medications, vitamins, or dietary supplements within 7 days of administration of the first dose of IMP, unless prior approval is granted by both the Principal Investigator and the Medical Monitor. Excluded from this list is intermittent use of acetaminophen £2 g/day or ibuprofen £1200 mg/day. Herbal supplements must be discontinued 14 days prior to the first dose of IMP.
15. Use of any antihistamines and/or decongestants within 30 days or nasal corticosteroids within 3 months prior to the first dose of IMP.
16. Consumed alcohol within 72 hours of Day -1 or have a positive alcohol test at Screening or admission to the CRU.
17. Subjects who consumed grapefruit juice or juices containing grapefruit or ate grapefruit or ate Seville oranges within 7 days prior to the first dose of IMP.
18. Excessive intake of caffeine-containing foods or beverages (more than 5 units or equivalent per day) within 48 hours prior to the admission to the study center (Day 1). One caffeine unit is contained in the following items: 1 (6 oz) cup of coffee, 2 (12 oz) cans of cola, 1 (12 oz) glass of tea, ½ (4 oz) cup of energy drink (e.g., Red Bull) or 3 (1 oz) chocolate bars.
19. Positive serum pregnancy test at the Screening Visit or positive urine pregnancy test on Day 1 (females only).
20. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (anti-HCV) at the Screening Visit.
21. Positive urine drug test at the Screening Visit or at admission to the CRU.
22. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.
23. Subjects who have donated blood or experienced other significant blood loss within 56 days of screening for the study.
24. Subjects with hemoglobin (Hb) <11 g/dL

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in adverse events from Baseline | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States